CLINICAL TRIAL: NCT06943482
Title: A Pilot Open-label Randomised Trial Comparing the Effectiveness of Steroids and Methotrexate for the Treatment of Idiopathic Granulomatous Mastitis
Brief Title: Comparing Effectiveness of Steroids and Methotrexate in Treatment of Chronic Inflammatory Breast Disease
Acronym: IGM
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/00773
Record Dates: First submitted 2025-03-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-11

CONDITIONS: Idiopathic Granulomatous Mastitis
Keywords: Breast; Breast Conditions; Mastits; Granulomatous Mastitis; Inflammation; Breast Surgery; Rhematologist
MeSH Terms: conditions — Granulomatous Mastitis; Inflammation | interventions — Prednisolone; Methotrexate; Folic Acid; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Steroid (Active Comparator)
  Interventions: Drug: Prednisolone; Drug: Omeprazole 20 mg
- Methotrexate (Experimental)
  Interventions: Drug: Methotrexate; Drug: Folic Acid 5 MG

INTERVENTIONS:
Drug: Prednisolone — 20mg of prednisolone will be prescribed, taken orally, and daily for first month followed by tapering doses of 15mg over one month, then 12.5mg for one month, proceeding to 10mg for one month, subsequently taking 7.5mg for one month, and lastly 5mg for one month.
  Arms: Steroid
Drug: Methotrexate — 10mg of methotrexate will be prescribed to be taken once a week for one month. The dosage will be increased to 15mg of methotrexate taken once a week on the 1st (T1) month clinical visit and will be further increased to 20mg of methotrexate taken once a week on the 2nd (T2) month clinical visit. There will be no further escalation of dosage after this visit.
  Arms: Methotrexate
Drug: Folic Acid 5 MG — 5mg of folic acid is to be taken together with methotrexate once a week.
  Arms: Methotrexate
Drug: Omeprazole 20 mg — Omeprazole will be prescribed at 20mg to protect the stomach lining.
  Arms: Steroid

SUMMARY:
This research study is to determine the effectiveness of prednisolone and methotrexate for IGM patients over a period of one year, in terms of clinical and radiological response. Recruitment will be conducted in National University Hospital (NUH) for patients diagnosed with IGM.

ELIGIBILITY:
Inclusion Criteria:

* Women, aged between 21 and 60 years
* Positive diagnosis of idiopathic granulomatous mastitis based on histopathology results
* Willing and able to give informed consent

Exclusion Criteria (Patients who meet any of the following prerequisites will not be allowed to take part in this study):

* Women who are currently pregnant or breastfeeding
* Cognitive impairment which prevents the patient from giving voluntary consent
* History of any psychiatric conditions such as depression, psychosis, schizophrenia etc.
* History of cancer in the past 5 years
* History of abnormal renal or liver function
* History of diabetes mellitus
* History of pulmonary lung disease, pneumonitis, or related conditions
* Hepatitis B and/or Hepatitis C carrier
* Diagnosed with tuberculosis (Positive microbiological evaluation for Grocott Methenamine Silver stain and Ziehl- Neelsen stain)
* Any immunosuppressants or anti-inflammatory medications such as NSAIDS for the past 3 months
* Concomitant medication that may have contraindication with prednisolone and methotrexate use
* Hypersensitivity to components or drug products of prednisolone and methotrexate
* Vaccination with live virus vaccines prior to or during treatment

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieved clinical or radiological complete response by 6 months | 6 months
Time to clinical response and time to radiological response | 6 months
Proportion of patients with relapse in a year within affected breast between each arm. | 1 year

SECONDARY OUTCOMES:
Evaluation of side effects. | 1 year
Evaluation of of treatment failure (TF) rate | 6 months
Evaluation of frequency of percutaneous or surgical intervention required | 6 months
Evaluation of potential unique pattern of gene expression that can be used to diagnose IGM and predict treatment response | 3 years
Evaluation of potential biomarkers that may predict response to treatment: eg IL-6, CRP and neutrophil to lymphocyte ratio (NLR) | 3 years
  Depending on the biomarkers tested, there will be different unit of measurements. Some examples of biomarkers that may be tested are:
  CRP: mg/l IL-6: pg/ml NLR: ratio
Evaluation of patient reported outcome measures | 3 years
  Most of our questions are on a scale from 1 - 5, with some yes or no question and an open question at the end.
Validate survey instrument for IGM patients | 3 years
  The survey is adopted from SF-36 for general health and EORTC BR23 for body image, breast health and pain.

CONTACTS AND LOCATIONS:
Overall Officials: Serene Si Ning Goh, MBBS, Principal Investigator — National
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altintoprak F, Kivilcim T, Ozkan OV. Aetiology of idiopathic granulomatous mastitis. World J Clin Cases. 2014 Dec 16;2(12):852-8. doi: 10.12998/wjcc.v2.i12.852. PMID 25516860
- [Background] Manogna, P., Dev, B., Joseph, L.D. et al. Idiopathic granulomatous mastitis-our experience. Egypt J Radiol Nucl Med 51, 15 (2020). https://doi.org/10.1186/s43055-019-0126-4
- [Background] Kehribar, D. Y., Duran, T. I., Cetinkaya, G. K., Polat, A. K., Ozgen, M. (2020). Evaluation of Symptoms, Depression and Anxiety Levels in Young Women with Idiopathic Granulomatous Mastitis. Int J Acad Med Pharm, 2(2), 57-61. https://doi.org/10.29228/jamp.42734
- [Background] Steuer AB, Stern MJ, Cobos G, Castilla C, Joseph KA, Pomeranz MK, Femia AN. Clinical Characteristics and Medical Management of Idiopathic Granulomatous Mastitis. JAMA Dermatol. 2020 Apr 1;156(4):460-464. doi: 10.1001/jamadermatol.2019.4516. PMID 31968055
- [Background] Al Awfi MM, Al Rahbi SK. Idiopathic Granulomatous Mastitis: Six years of experience and the current evidence in literature. Sultan Qaboos Univ Med J. 2023 Feb;23(1):36-41. doi: 10.18295/squmj.4.2022.030. Epub 2023 Feb 23. PMID 36865415
- [Background] Kayahan M, Kadioglu H, Muslumanoglu M. Management of Patients with Granulomatous Mastitis: Analysis of 31 Cases. Breast Care (Basel). 2012 Jun;7(3):226-230. doi: 10.1159/000337758. Epub 2012 Jun 27. PMID 22872797
- [Background] Kafadar MT, Bahadir MV, Girgin S. Low-Dose Methotrexate Use in Idiopathic Granulomatous Mastitis: An Alternative Treatment Method. Breast Care (Basel). 2021 Aug;16(4):402-407. doi: 10.1159/000513879. Epub 2021 Jan 22. PMID 34602947
- [Background] Kim J, Tymms KE, Buckingham JM. Methotrexate in the management of granulomatous mastitis. ANZ J Surg. 2003 Apr;73(4):247-9. doi: 10.1046/j.1445-1433.2002.02564.x. PMID 12662235
- [Background] Postolova A, Troxell ML, Wapnir IL, Genovese MC. Methotrexate in the Treatment of Idiopathic Granulomatous Mastitis. J Rheumatol. 2020 Jun 1;47(6):924-927. doi: 10.3899/jrheum.181205. Epub 2019 Jun 15. PMID 31203215
- [Background] Sheybani F, Sarvghad M, Naderi H, Gharib M. Treatment for and clinical characteristics of granulomatous mastitis. Obstet Gynecol. 2015 Apr;125(4):801-807. doi: 10.1097/AOG.0000000000000734. PMID 25751209